CLINICAL TRIAL: NCT02990065
Title: Optimizing Protein Intake and Nitrogen Balance in Adult Critically Ill Patients: a Randomized Controlled Trial (OPINiB STUDY)
Brief Title: Optimizing Protein Intake and Nitrogen Balance in Adult Critically Ill Patients
Acronym: OPINiB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Dario Gregori, Associate Professor, University of Padova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OPINiB 2016
Record Dates: First submitted 2016-11-28; First posted 2016-12-12 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Protein Deficiency
Keywords: PROTEIN SUPPLEMENTATION; NUTRITIONAL STATUS
MeSH Terms: conditions — Protein Deficiency

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- PROTEIN-FORTIFIED DIET (Experimental): The protein-fortified diet consists on an energy goal based on REE measurement and a protein target based on the most recent literature recommendations (1.2-2 g/kg/die) (2). Daily caloric requirement, and subsequent protein content, of patients enrolled in the intervention group will be calculated using formulas in Table 1 (10, 12, 13). For each patient will be calculated the Resting Energy Expenditure (REE) and daily protein requirement (1.2-2g/kg/die of body weight registered at the admission) and the corresponding caloric intake (1g = 4 kcal). Finally, total daily caloric intake will be calculated by adding kcal from protein (1g = 4kcal) on kcal from non-protein (50% of REE).
  Interventions: Dietary Supplement: PROTEIN SUPPLEMENTATION
- STANDARD DIET (No Intervention): The standard diet consists on an energy goal based on weight formula (20-25 kcal/kg/die). According to the ICU nutritional protocol, EN is started at an initial rate of 10ml/h, and increased by 20ml/h every 12 hours in the absence of significant gastric residuals (<250ml), with the aim of reaching the energy goal within 72 hours from admission. The EN formulae used are standard (1-1,5 kcal/ml, 40g/l protein). If enteral nutrition is not tolerated or is not indicated, supplemental PN is used to make up the energy shortfall. The PN formula used is standard (1000 kcal/l, 37 g/l protein).

INTERVENTIONS:
Dietary Supplement: PROTEIN SUPPLEMENTATION
  Arms: PROTEIN-FORTIFIED DIET

SUMMARY:
The purposes of the study are:

* To strictly ensure the appropriate level of protein and caloric provision in critical illness, according to the latest literature recommendation;
* To determine if an association exists between protein intake and nitrogen balance in the context of a nutrition with appropriate protein provision based on the latest literature recommendations, rather than in a standard diet with a caloric target weight-based. Creatinine clearance will also be evaluated to determine if there is any harmful effect to the kidney secondary to an elevated BUN.
* To determine if there is a difference in ICU mortality rate between the current nutrition standard and a hyperproteic nutrition protocol.

ELIGIBILITY:
Inclusion criteria:

* Age > 18 years
* Receiving PN and/or EN nutrition
* Indwelling urinary catheter
* Mechanically ventilated patients

Exclusion criteria:

* Age < 18 years
* Chronic renal or hepatic failure
* Current or history (past 6 months) of GI bleeding
* BMI >30 kg/m2 o <18 kg/m2
* Terminally ill patients
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
nitrogen balance (gr) | change from baseline through study completion, an average of 15 days
  (gr)

REFERENCES:
- [Derived] Danielis M, Lorenzoni G, Cavaliere L, Ruffolo M, Peressoni L, De Monte A, Muzzi R, Beltrame F, Gregori D. Optimizing Protein Intake and Nitrogen Balance (OPINiB) in Adult Critically Ill Patients: A Study Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2017 May 9;6(5):e78. doi: 10.2196/resprot.7100. PMID 28487264